CLINICAL TRIAL: NCT07395089
Title: Atrial Remodeling Associated With Pulse-Field Ablation of Atrial Fibrillation: a Computed Tomography Study
Brief Title: Computed Tomography of Pulse-Field Ablation
Acronym: CT-PFA
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: NIXXXXXHLJ
Record Dates: First submitted 2025-11-28; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-02

CONDITIONS: Atrial Fibrillation (AF); Arrhythmia
Keywords: Ablation; Reverse Atrial Remodeling; Radiofrequency Catheter Ablation; Pulse Field Ablation; Pulmonary Vein Reconnexion; Epicardial Adipose Tissue
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pulse-Field Ablation
- Radiofrequency Catheter Ablation

SUMMARY:
Radiofrequency catheter ablation (RFCA) of atrial fibrillation (AF) reduces left atrial (LA) volume post-ablation, a phenomenon termed reverse atrial remodeling, indicative of successful reversal of atrial cardiomyopathy progression. In contrast, pulse field ablation (PFA), a novel non-thermal technology, offers a promising efficacy and safety profile without inducing persistent atrial fibrosis. While RFCA-associated reverse atrial remodeling is well-documented, it remains uncertain whether PFA, operating on a non-thermal paradigm, also promotes this remodeling, which would enhance its physiological relevance in AF treatment. Additionally, RFCA studies show that LA wall thickness at the pulmonary vein (PV) antrum can predict PV reconnection and arrhythmia recurrence, but whether PFA affects LA thinning or enables similar predictions from post-treatment computed tomography (CT) scans is unknown. Moreover, epicardial adipose tissue (EAT), strongly linked to LA abnormalities and AF recurrence, can be quantified via CT, yet the impact of PFA on LA EAT remains unexplored. Finally, PFA's versatility, particularly in isolating the LA posterior wall (LAPW) in non-paroxysmal AF, raises questions about its effect on posterior wall thinning or EAT changes, factors associated with post-ablation recurrence

ELIGIBILITY:
Inclusion Criteria:

1. Age≥18 years at the time of AF ablation
2. AF ablation by pulse-field ablation (BOSTON SCIENTIFIC FARAPULSE) or by radiofrequency (any manufacturer) between 2020 and 2024
3. Paroxysmal or non-paroxysmal AF
4. Pre-ablation CT data available and of high quality
5. Post-ablation CT data available and of high quality
6. Post-ablation CT performed 3-months (+- 2 weeks) after AF ablation

Exclusion Criteria:

1. Low quality CT, non-homogeneous contrast agent perfusion
2. Post-ablation CT performed in another center
3. Patients in which pre- and post-ablation CTs do not share common phases
4. Patients who underwent ethanol infusion in the vein of Marshall

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients at Hôpital Pitié Salpêtrière meeting the study criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Difference between baseline and post-ablation LA indexed volume (ml/cm^2) | Post-procedural (3-months)

SECONDARY OUTCOMES:
Difference between baseline and post-ablation mean wall thickness, mm | Post-procedural (3-months)
Difference between baseline and post-ablation Epicardial adipose tissue , mm^3 | Post-procedural (3-months)
Difference between baseline and post-ablation left atrial appendage indexed volume, ml/cm^2 | Post-procedural (3-months)
Difference between baseline and post-ablation left atrial appendage dimensions (long-axis, short-axis, ostium long-axis, ostium short-axis), mm | Post-procedural (3-months)
Difference between baseline and post-ablation mean LA wall thickness at the LAPW, mm | Post-procedural (3-months)
Difference between baseline and post-ablation epicardial adipose tissue at the PW, mm^3 | Post-procedural (3-months)
Recurrence of sustained atrial arrhythmia | Post-procedural (3-months)
Recurrence of sustained atrial arrhythmia | 12 months after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Carine Paré, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié Salpêtrière, Paris, Île-de-France Region, France